CLINICAL TRIAL: NCT01217164
Title: Strategy to Minimize In-hospital Malnutrition in Premature Babies
Acronym: SPN
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hospital Universitario Pedro Ernesto (Other)
Responsible Party: Jose Luiz Muniz Bandeira Duarte, Faculdade de Ciencias Médicas, UERJ
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DUARTEJLMB-001
Record Dates: First submitted 2010-08-27; First posted 2010-10-08 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Weight Gain Preterm
Keywords: nutrition; very low birth weight; premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- higher protein (No Intervention)
  Interventions: Dietary Supplement: no intervention

INTERVENTIONS:
Dietary Supplement: no intervention — received enteral diet with 4.5 g / kg / day of protein and 160cal/Kg/dia
  Other Names: Feeding preterm; Very low birth weight; weight gain; neurodevelopment

SUMMARY:
Adequate nutrition is important for preventing malnutrition in the postnatal period and thus optimize growth and development of children born prematurely. To avoid malnutrition is recommended to provide nutrients necessary for a growth rate similar to the intrauterine life.

For nearly one decade studying how to minimize in-hospital malnutrition in children born prematurely, especially with gestational age less than 32 weeks or with birth weight below 1,500 g, called newborn very low birth weight (VLBW).

Embleton et al.demonstrated that with the current nutritional recommendations (protein between 3.0 and 3.8 g / kg / day), the VLBW had malnutrition caused by protein and calorie cumulative deficit.

Poor nutrition in the neonatal period can impair growth and neuromotor and cognitive development after hospital discharge.

The investigators hypothesis is that VLBW subjected to aggressive nutrition with protein-calorie high from birth until discharge, would present higher weight gain than the VLBW infants who received routine diet of service, without producing adverse effects.

DETAILED DESCRIPTION:
The study used newborn with weight less than or equal to 1,500, at the University Hospital Pedro Ernesto (HUPE) State University of Rio de Janeiro. Were defined as exclusion criteria congenital malformations, genetic syndromes and death of the patient before inclusion in the study. All children included in the study after written consent of those responsible, received aggressive parenteral nutrition immediately after birth and minimal enteral feeding in the first or second day of life. When the volume of enteral diet reached the value equal to or greater than 100 ml / kg / day was suspended intravenous hydration or parenteral nutrition. The increase of enteral nutrition was conducted in compliance with the gradual increase of 20 ml / kg / day, according the acceptance of VLBW.The clinical trial was randomized into two types of calorie intake in the diet. Newborn exposed group (EG) received enteral diet with 4.5 g / kg / day of protein and 160cal/Kg/dia, and in the control group (CG) was used usual diet with caloric intake from 3.5 to 4 g / kg / day of protein and 120-140 kcal / kg / day. The osmolality of the diet has not changed, there was an increase in the volume to achieve the desired protein-caloric. We used two types of nutrition: 1) raw milk milked exclusively at the bedside of VLBW (without fortifying additive); 2) milk formula for premature exclusive. The type of feed was considered as exclusive breastfeeding or exclusive formula for premature when there were more than 80% predominance of one type of food. The food was offered initially by orogastric catheter until the child reaches maturity to be fed by cup and / or suction.

The assessment was initiated when enteral feeding reached a volume exceeding 100 ml / kg / day and was suspended concomitant intravenous infusion or nutrition parenteral total (NPT) solution, and completed at discharge or at 43 weeks corrected gestational age, or in case of death or shutdown of the project requested by those responsible.

The calculation of caloric intake and water was daily, were presumed to breast milk values of 1.5 g of protein and 70 calorias/100 ml and in milk formula for premature infants used are listed values of 2.3 g of protein and 80 calories per 100ml.The outcome measure will be assessed when children have completed 43 weeks of corrected gestational age.

The sample size calculation assuming risk of 5%, 80% power and prevalence of 50% resulted in 60 newborn. Statistical analysis were measured average rates of weight and gestational age at birth and at discharge, the average corrected age at discharge, the rate of SGA VLBW; daily weight gain during the total days of hospitalization, the real weight gain during the period between the day of recovery of birth weight and hospital discharge. Was also calculated the difference between Z score of hospital discharge and birth for weight, length and head circumference.

Statistical calculations were performed: Ficher exact test and / or odds ratio (OR) for categorical variables, ANOVA or Kruskal-Wallis test for continuous variables. Was considered when p <0.05 as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All very low birth weight infant after written consent of those responsible

Exclusion Criteria:

* congenital malformations, genetic syndromes and death

Max Age: 43 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2008-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The total of 64 children was followed from birth until discharge or death. The main outcome measured was weight gain during hospitalization or up to a maximum of 43 weeks gestational age when the child remained hospitalized | The cutoff point for the measurement of weight was discharged or until 43 weeks corrected gestational age if prolonged hospitalization.
  The results measured were: 1- the real gain in weight (weight gain during hospitalization days divided by the number of days between birth weight recovery until discharge day or time he turned 43 weeks corrected gestational age). 2 - The weight gain during hospitalization (weight gain during hospitalization divided by the number of days between the day of birth until the day of discharge).

SECONDARY OUTCOMES:
The difference between score Z (birth weight) and score Z (weight during discharge). | The cutoff point for the measurement of weight was discharged or until 43 weeks corrected gestational age if prolonged hospitalization.
  Measurements of the Z score corresponding to the birth weight and weight were discharged through the growth curve of the WHO (2006)

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Duarte, Principal Investigator — State University of Rio de Janeiro
Locations (1):
- Jose Luiz Muniz Bandeira Duarte, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Result] Ehrenkranz RA, Younes N, Lemons JA, Fanaroff AA, Donovan EF, Wright LL, Katsikiotis V, Tyson JE, Oh W, Shankaran S, Bauer CR, Korones SB, Stoll BJ, Stevenson DK, Papile LA. Longitudinal growth of hospitalized very low birth weight infants. Pediatrics. 1999 Aug;104(2 Pt 1):280-9. doi: 10.1542/peds.104.2.280. PMID 10429008
- See also: university hospital ou state university of rio de janeiro — http://www.hupe.uerj.br